CLINICAL TRIAL: NCT00147966
Title: Assessment of the Immunomodulatory Effects of Rituximab in Seropositive Rheumatoid Arthritis Using Arthroscopic Synovial Biopsies
Brief Title: Assessment of Rituximab's Immunomodulatory Synovial Effects (The ARISE Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Arthur Kavanaugh, UCSD
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 041569
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Results first posted 2010-03-23 (Estimated); Last update posted 2010-03-23 (Estimated); Status verified 2008-06

CONDITIONS: Rheumatoid Arthritis
Keywords: active disease despite concomitant methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ritxumab (Experimental): all patients get treatment
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab — treatment with rituximab
  Other Names: rituxan

SUMMARY:
Using repeated arthroscopic biopsies of patients with rheumatoid arthritis, the researchers will assess changes in the immune response that occur as a result of treatment with rituximab.

DETAILED DESCRIPTION:
Using repeated arthroscopic biopsies of patients with rheumatoid arthritis, the researchers will assess changes in the immune response that occur after treatment with rituximab.

ELIGIBILITY:
Inclusion Criteria:

* Active rheumatoid arthritis
* Use of concomitant methotrexate

Exclusion Criteria:

* Use of disease-modifying anti-rheumatic drugs (DMARDs)/biologics other than methotrexate
* Serious medical conditions that would preclude the use of the treating agent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Kavanaugh, MD, Principal Investigator — UCSD CIT
Locations (1):
- UCSD CIT, La Jolla, California, United States

REFERENCES:
- [Background] Kavanaugh A, Rosengren S, Lee SJ, Hammaker D, Firestein GS, Kalunian K, Wei N, Boyle DL. Assessment of rituximab's immunomodulatory synovial effects (ARISE trial). 1: clinical and synovial biomarker results. Ann Rheum Dis. 2008 Mar;67(3):402-8. doi: 10.1136/ard.2007.074229. Epub 2007 Jul 20. PMID 17644541
- [Background] Rosengren S, Wei N, Kalunian KC, Zvaifler NJ, Kavanaugh A, Boyle DL. Elevated autoantibody content in rheumatoid arthritis synovia with lymphoid aggregates and the effect of rituximab. Arthritis Res Ther. 2008;10(5):R105. doi: 10.1186/ar2497. Epub 2008 Sep 1. PMID 18761748
- [Derived] Rosengren S, Wei N, Kalunian KC, Kavanaugh A, Boyle DL. CXCL13: a novel biomarker of B-cell return following rituximab treatment and synovitis in patients with rheumatoid arthritis. Rheumatology (Oxford). 2011 Mar;50(3):603-10. doi: 10.1093/rheumatology/keq337. Epub 2010 Nov 23. PMID 21098574

RESULTS

PARTICIPANT FLOW:
Groups:
- Ritxumab: Rituximab at a dose of 1000 mg was given intravenously over 4-5 hours on day 0, and again on day 14.
Period: Overall Study
Arm/Group | Ritxumab
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ritxumab
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology (ACR) 20 at Week 12
Description: ACR 20, the American College of Rheumatology (ACR) definition of 20% improvement is based on a 20% improvement (compared to baseline values) in tender and swollen joint counts and 20% improvement in 3 of the remaining 5 core set measures (subject global assessment of pain, subject global assessment of disease activity, physician global assessment of disease activity, subject assessment of physical function) and one acute phase reactant value (CRP).
Time Frame: 0 and 12 weeks
Measure: Number; unit: participants
Arm/Group | Ritxumab
Number analyzed (Participants) | 24
participants | 12

ADVERSE EVENTS:
Arm/Group | Ritxumab
Serious Adverse Events (participants affected / at risk) | 2/24
Other Adverse Events (participants affected / at risk) | 21/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ritxumab (N=24)
Anemia (Blood and lymphatic system disorders) | 1 (1) — considered not related to study drug
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 1 (1) — considered not related to study drug
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — considered not related to treatment with study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ritxumab (N=24)
Allergic reaction to detergent on hand and arm (Immune system disorders) | 1
Hot/cold flashes (General disorders) | 1
Contact dimities (Skin and subcutaneous tissue disorders) | 1
Edema (Vascular disorders) | 1
Excessive vaginal bleeding (Reproductive system and breast disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Deep venous thrombosis (Vascular disorders) | 1
Leg small vessel bursting (Vascular disorders) | 1
Spider veins (Vascular disorders) | 1
Headache (Nervous system disorders) | 1
Sinus headache (Immune system disorders) | 1
Dizziness (Nervous system disorders) | 1
Fatigue (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Insomnia (Nervous system disorders) | 1
Hair loss (Skin and subcutaneous tissue disorders) | 1
Fall (General disorders) | 1
Lacerated forehead (Injury, poisoning and procedural complications) | 1
Hiatal hernia (Gastrointestinal disorders) | 1
Corrective surgery, hammer toes (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No